CLINICAL TRIAL: NCT02272998
Title: Phase II Study of Ponatinib for Advanced Cancers With Genomic Alterations in Fibroblastic Growth Factor Receptor (FGFR) and Other Genomic Targets (KIT, PDGFRá, RET FLT3, ABL1)
Brief Title: Ponatinib for Patients Whose Advanced Solid Tumor Cancer Has Activating Mutations Involving the Following Genes: FGFR1, FGFR2, FGFR3, FGFR4, RET, KIT.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sameek Roychowdhury (Other)
Responsible Party: Sponsor-Investigator, Sameek Roychowdhury, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-14078; NCI-2014-01499 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-10-21; First posted 2014-10-23 (Estimated); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Malignant Neoplasm
Keywords: FGFR, RET, KIT
MeSH Terms: conditions — Neoplasms; Piebaldism | interventions — ponatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ponatinib hydrochloride) (Experimental): Patients receive ponatinib hydrochloride PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: ponatinib hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: ponatinib hydrochloride — Given PO
  Other Names: AP24534; Iclusig; multitargeted tyrosine kinase inhibitor AP24534
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well ponatinib hydrochloride works in treating patients with cancer that has spread to other parts of the body (metastatic), has failed previous treatment (refractory), and has one of several alterations, or mutations, in its deoxyribonucleic acid (DNA) sequence. Ponatinib hydrochloride may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. It is not yet known whether a patient's genetic alterations may affect how well ponatinib hydrochloride works.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the response of ponatinib (ponatinib hydrochloride) in patients with fibroblast growth factor receptor (FGFR) altered cancers.

SECONDARY OBJECTIVES:

I. To assess the safety and tolerability of ponatinib in advanced solid tumors with genomic FGFR alterations.

II. To assess progression free survival (PFS) and overall survival (OS) with ponatinib.

III. To determine candidate genomic and proteomic biomarkers of sensitivity and resistance to ponatinib using unbiased high throughput approaches (exome, transcriptome, reverse phase protein array [RPPA]).

IV. To assess response of ponatinib in advanced cancers with subsets of genomic FGFR alterations (fusions vs. amplifications vs. mutations).

OUTLINE:

Patients receive ponatinib hydrochloride orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed diagnosis of refractory metastatic solid tumor or chronic hematological malignancy who are eligible for investigational drug therapy
* Patients must have tumor suitable for biopsy (as assessed by trained specialists in interventional radiology) and medically fit to undergo a biopsy or surgical procedure OR if patients do not have a tumor suitable for biopsy but have another tissue available for molecular evaluation
* Patients should have activating genomic alterations in FGFR (mutations, fusions or amplifications [> 6 copies]) or activating genomic alterations in KIT, platelet-derived growth factor receptor alpha [PDGFRα], ret proto-oncogene [RET], ABL proto-oncogene 1, non-receptor tyrosine kinase [ABL1] and fms-related tyrosine kinase 3 [FLT3] by any validated Clinical Laboratory Improvement Amendments [CLIA]-certified molecular testing (fluorescent in situ hybridization [FISH], polymerase chain reaction [PCR] or sequencing data are acceptable); CLIA validated results from other institutions; diagnostic labs (e.g. foundation medicine) are acceptable; additional types of activating alterations in these genes can be approved by the principal investigator (PI)
* Patients with advanced cancers should have had at least one prior therapy that is considered standard for that disease type
* Patients with solid tumors must have measurable disease (Response Evaluation Criteria in Solid Tumors [RECIST] 1.1), defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 80%)
* Life expectancy of greater than 3 months
* Patients with multiple malignancies remain eligible
* Patients with an inherited cancer syndrome or a medical history suggestive of an inherited cancer syndrome remain eligible
* Patients must have controlled blood pressure with a systolic blood pressure < 140 mmHg and diastolic < 90 mmHg; anti-hypertensive medications are permitted
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and through 4 months after the end of treatment; for females of childbearing potential, a negative pregnancy test must be documented prior to randomization
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 75,000/mcL
* Total bilirubin =< 1.5 x upper limit of normal (ULN), unless due to Gilbert's syndrome (< 5 if liver involvement with primary tumor)
* Serum lipase and amylase =< 1.5 x ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Left ventricular ejection fraction (LVEF) >= institutional lower limit of normal by echocardiogram (ECHO) or multi gated acquisition (MUGA)
* Serum creatinine =< 1.5 mg/dL OR calculated creatinine clearance (Cockcroft-Gault formula) >= 50 mL/min OR 24-hour urine creatinine clearance >= 50 mL/min
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with acute hematological malignancies
* Patients who have not received any prior treatment.
* Patients with known ponatinib-resistant gene alterations

  * PDGFRA D842V mutation
  * cKIT D816V mutation
  * FLT3 D835V/Y/H/F or Y842C mutations
  * FGFR3 K652E mutation
* Major surgery (e.g. thoracic, abdominal, vascular, neurosurgery) within 28 days prior to initiating therapy
* History of acute pancreatitis within one year of study or history of chronic pancreatitis
* History of alcohol abuse
* Have uncontrolled hypertriglyceridemia (triglycerides > 450 mg/dL)
* Patients with history of clinically significant bleeding disorder
* Pregnant women are excluded from this study because ponatinib can affect embryo-fetal development. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ponatinib breastfeeding must be discontinued.
* Patients who are incarcerated are not eligible
* Patients with any history of arterial thromboembolic disease; any patient with a history of myocardial infarction (MI), stroke, transient ischemic attack (TIA), unstable angina or peripheral vascular disease will not be eligible
* Patients with history of recurrent venous thromboembolism (deep venous thrombosis or pulmonary embolism) or history of venous thromboembolism within 6 months will not be eligible
* Patients with history of active hepatitis B or C infection or chronic hepatitis with Child Pugh B or C hepatic dysfunction
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ponatinib
* Patients with prolonged corrected QT interval, defined as QTc >450 msec
* Use of antiplatelet agents other than low-dose aspirin as described
* GI bleed within 30 days prior to registration on study
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ponatinib.
* Patients with history of atrial arrhythmia (requiring any anti-arrhythmic therapy) or patients with any history of ventricular arrhythmia are excluded
* Clinically significant, uncontrolled intercurrent illness including, but not limited to:

  * Symptomatic or active infection
  * Uncontrolled hypertension (diastolic blood pressure > 90 mm Hg; systolic > 140 mm Hg); patients with hypertension should be under treatment on study entry to effect blood pressure control
  * Psychiatric illness/social situations that would limit compliance with study requirements
* Patients with history of congestive heart failure are excluded
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with ponatinib.
* Patients on medications known to be associated with Torsades de Pointes
* Patients who received the last administration of an anti-cancer therapy including, chemotherapy, immunotherapy/biologic therapy, targeted therapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) or within 5 half-lives, whichever is shorter, prior to entering the study.
* Patients taking medications or herbal supplements that are known to be strong cytochrome P450 3A4 (CYP3A4) inhibitors within at least 14 days before the first dose of ponatinib are excluded
* Patients with symptomatic or progressive brain metastases are ineligible; subjects with treated brain metastases are eligible if they have no radiographic or other signs of progression in the brain for >= 4 weeks after completion of local therapy
* Patients with macular edema, retinal vein occlusion or retinal hemorrhage are excluded.
* Patients who have received prior FGFR targeted therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-02-24 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sameek Roychowdhury, MD, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Ponatinib Hydrochloride)
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ponatinib Hydrochloride)
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Overall Response, Defined as the Number of Patients Who Achieve Any Response According to Disease Type in the First 6 Courses of Treatment
Description: The proportion of responses for the purposes of the decision rule will be calculated out of all eligible patients who receive any treatment. Assuming the number of responses is binomially distributed, 95% binomial confidence intervals will also be calculated for the estimate of the proportion of responses. Response for tumors was assessed using the RECIST 1.1 criteria (using computed tomography [CT] scans), where response was defined as a partial or complete response.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Participants With Genomic Alterations in FGFR; Participants With Genomic Alterations in Rare Genomic Targets (KIT, PDGFRα, RET, ABL1, and FLT3): Patients receive ponatinib hydrochloride PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  ponatinib hydrochloride: Given PO
  laboratory biomarker analysis: Correlative studies
Arm/Group | Participants With Genomic Alterations in FGFR | Participants With Genomic Alterations in Rare Genomic Targets (KIT, PDGFRα, RET, ABL1, and FLT3)
Number analyzed (Participants) | 17 | 5
Participants | 1 | 0

2. Secondary Outcome: Percentage of Participants With Adverse Events, Defined as Adverse Events That Are Classified as Either Possibly, Probably, or Definitely Related to Study Treatment Per National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: Frequency and severity of adverse events will be collected and summarized by descriptive statistics. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns for each of the cohorts as well as across cohorts. In addition, all adverse event data that is graded as 3, 4, or 5 will be reviewed and classified as either "unrelated" or "unlikely to be related" to study treatment in the event of an actual relationship developing.
Time Frame: Up to 30 days after last dose of study drug, up to a total of 6 years
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Ponatinib Hydrochloride)
Number analyzed (Participants) | 22
percentage of participants
  Dry Skin, Grade 1 | 36.4
  Dry Skin, Grade 2 | 4.6
  Dry Skin, Grade ≥3 | 9.1
  Rash Maculo-papular, Grade 1 | 27.3
  Rash Maculo-papular, Grade 2 | 9.1
  Hypertension, Grade 1 | 4.6
  Hypertension, Grade 2 | 9.1
  Hypertension, Grade ≥3 | 13.6
  Fever, Grade 1 | 27.3
  Alkaline Phosphatase Increased, Grade 1 | 4.6
  Alkaline Phosphatase Increased, Grade 2 | 13.6
  Alkaline Phosphatase Increased, Grade ≥3 | 4.6
  Headache, Grade 1 | 13.6
  Headache, Grade 2 | 9.1
  Nausea, Grade 1 | 9.1
  Nausea, Grade 2 | 9.1
  Abdominal Pain, Grade ≥3 | 13.6
  Lymphocyte Count Decreased, Grade 1 | 4.6
  Lymphocyte Count Decreased, Grade 2 | 4.6
  Lymphocyte Count Decreased, Grade ≥3 | 4.6
  Anorexia, Grade 1 | 4.6
  Anorexia, Grade 2 | 9.1
  Alanine Aminotransferase Increased, Grade 1 | 13.6
  Fatigue, Grade 1 | 9.1
  Fatigue, Grade 2 | 4.6
  Pancreatitis, Grade 2 | 4.6
  Pancreatitis, Grade ≥3 | 4.6
  Dyspnea, Grade 2 | 4.6
  Dyspnea, Grade ≥3 | 4.6
  Dry Mouth, Grade 1 | 9.1
  Mucositis, Grade 1 | 9.1
  Diarrhea, Grade 1 | 9.1
  Aspartate Aminotransferase Increased, Grade 1 | 9.1
  Dysgeusia, Grade 1 | 4.6
  Dysgeusia, Grade 2 | 4.6
  Arthralgia, Grade 1 | 4.6
  Arthralgia, Grade 2 | 4.6
  Serum Amylase Increased, Grade ≥3 | 4.6
  Supraventricular Tachycardia, Grade ≥3 | 4.6
  Lipase Increased, Grade ≥3 | 4.6
  Palmar-plantar Erythrodysesthesia Syndrome, Grade 1 | 4.6
  Thromboembolic Event, Grade 2 | 4.6

3. Secondary Outcome: Tolerability of the Regimen, Assessed by the Number of Patients Who Required Dose Modifications and/or Dose Delays
Description: Collected and summarized by descriptive statistics.
Time Frame: Up to 30 days after last dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ponatinib Hydrochloride)
Number analyzed (Participants) | 22
Participants | 11

4. Secondary Outcome: Overall Survival
Description: Kaplan-Meier curves will be used to estimate the survival distribution.
Time Frame: The time from treatment initiation to death, assessed up to 72 months
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Ponatinib Hydrochloride)
Number analyzed (Participants) | 22
months | 5.3 [0 to 72]

5. Secondary Outcome: Progression Free Survival
Description: Kaplan-Meier curves will be used to estimate the survival distribution.
Time Frame: The time from treatment initiation to progression or death, assessed up to 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Ponatinib Hydrochloride)
Number analyzed (Participants) | 22
months | 1.9 [0 to 19.7]

6. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Calculated by the number of patients who have achieve a response and/or are progression-free and alive at 6 months divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for CBR will be calculated.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Ponatinib Hydrochloride)
Number analyzed (Participants) | 22
percentage of participants | 31.8

7. Other Pre Specified Outcome: Correlative Gene and Protein Markers
Description: Correlative gene and protein markers will be summarized univariately in a quantitative manner and also summarized by clinical outcome group (e.g. response vs. no response). Graphical analyses will be largely used to assess potential patterns and relationships; e.g. side-by-side boxplots to assess differences in continuous marker levels between those with vs. without the clinical improvement (e.g. response vs. no response). Overall, hypothesis testing will largely be avoided given the sample size limitations.
Time Frame: Up to 3 years (time of progression)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each patient from the start of treatment with the investigational drug up to 30 days after ending treatment. The total time period in which adverse event data was collected for this study was 6 years.
Arm/Group | Treatment (Ponatinib Hydrochloride)
All-Cause Mortality (participants affected / at risk) | 16/22
Serious Adverse Events (participants affected / at risk) | 3/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ponatinib Hydrochloride) (N=22)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Thromboembolic Event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ponatinib Hydrochloride) (N=22)
Abdominal cramping (Gastrointestinal disorders) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 8 (8)
Alanine aminotransferase increased (Investigations) | 3 (3)
Alanine transaminase increased (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 7 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 12 (12)
Anorexia (Metabolism and nutrition disorders) | 12 (12)
Anxiety (Psychiatric disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9)
Breast pain (Reproductive system and breast disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 4 (4)
Confusion (Psychiatric disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 15 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Creatinine increased (Investigations) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Depression (Psychiatric disorders) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 9 (9)
Dizziness (Nervous system disorders) | 3 (3)
Dry eye (Eye disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 6 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 15 (15)
Dysesthesia (Nervous system disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 (14)
Dysuria (Renal and urinary disorders) | 2 (2)
Edema limbs (General disorders) | 7 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Eye disorders, other (Eye disorders) | 5 (5)
Fatigue (General disorders) | 20 (20)
Fever (General disorders) | 9 (9)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Flushing (Vascular disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Glucose Intolerance (Metabolism and nutrition disorders) | 3 (3)
Headache (Nervous system disorders) | 8 (8)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (8)
Hypertension (Vascular disorders) | 9 (9)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (5)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 7 (7)
Itching (Skin and subcutaneous tissue disorders) | 2 (2)
Lymphocyte count decreased (Investigations) | 7 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 (9)
Mucositis oral (Gastrointestinal disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 13 (13)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Pancreatic Enzymes Decreased (Investigations) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 3 (3)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (6)
Weight Loss (Investigations) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/98/NCT02272998/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/98/NCT02272998/ICF_001.pdf